CLINICAL TRIAL: NCT06638684
Title: Effects of High- and Moderate-intensity Exercise on T Cell Function in Healthy Young Men
Brief Title: T Cell Responses to Various Levels of Exercise Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas (Other)
Responsible Party: Principal Investigator, Philip Gallagher, Professor, University of Kansas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00001969; ONR N000141410202 (Other Grant/Funding Number: Office of Navel Research)
Record Dates: First submitted 2024-10-03; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Healthy
Keywords: Immune; Cytokine; Flow Cytometry; Immunoendocrine
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Moderate intensity exercise (Active Comparator): Subjects will participate in a 100 min bout of exercise led by an exercise physiologist doing the same exercises as the high-intensity group, but at a lower effort level. Exercise consists of of a mix of running activities (≤ 400 m); body weight exercises, such as burpees and lunges; and exercises, such as crunches and squats utilizing 20.4 kg weight plates, but performed at a pace allowing for in-session recovery. Scheduled 5 min rests will be included at 30, 60, and 85 min and MI subjects will be similarly encouraged to consume water and/or the carbohydrate/electrolyte drink. The researchers will obtain a blood sample from you prior to and immediately following the exercise, as well as one, four and six hours post-exercise.
  Interventions: Other: Exercise
- High intensity exercise (Experimental): Subjects in this group will participate in an exercise session that is representative of a training event experienced by cadets preparing for military competitions. All exercises will consist of a mix of running activities (≤ 400 m); body weight exercises, such as burpees and lunges; and exercises, such as crunches and squats utilizing 20.4 kg weight plates; with rapidly occurring exercise transitions to prevent recovery. The exercise bout will last a total of 100 min. Scheduled 5 min rests will be inserted at 30, 60, and 85 min. During the scheduled rest periods, subjects will be encouraged to consume water and/or the carbohydrate/electrolyte drink. The researchers will obtain a blood sample from you prior to and immediately following the exercise, as well as one, four and six hours post-exercise.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Subjects in the two groups preformed 90-100 minutes of exercise at different intensities.
  Other Names: Moderate-intensity; High-intensity

SUMMARY:
The objective of this project is to quantify the immunoendocrine response to acute stress events combining both physical and psychological challenges. This work will serve as a pilot project examining differential stress induction in response to exercise. Participants will have an instructor with prior military training lead a two-hour training session for 10 recreationally fit male volunteers. You will be randomly assigned to a high-intensity training group to participate in the "military style" training and a low-intensity training group who will participate in a low-intensity cardiovascular training protocol. Blood samples will be collected from you prior to and following the exercise session and these samples will be analyzed for endocrine measures as well as markers of immune function to include chemokines and cytokines.

ELIGIBILITY:
All subjects will be screened using a health-history questionnaire for contradictions to exercise by American College of Sports Medicine (ACSM) guidelines

Inclusion Criteria:

* Recreationally active
* Between the ages of 18-40,
* Healthy
* Non-obese (BMI <28 kg/m2)
* Non-smoking
* Free of metabolic or cardiovascular diseases.

Exclusion Criteria:

* Unhealed Fractures
* Thrombophlebitis (blood clots)
* Recent Surgery (within the last three months)
* Recent Uncontrolled Bruising
* Osteomyelitis (acute or chronic bone infection)
* Myositis Ossificans (hardened scarring in muscle tissue of the thigh).

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-02-20 (Actual); Primary Completion 2016-05-12 (Actual); Study Completion 2016-05-12 (Actual)

PRIMARY OUTCOMES:
T cell proliferation | 6.5 hours
  Blood samples were collected using standard venipuncture technique. Blood samples were obtained at baseline, immediately post-exercise (0h), 1 hour post (1h), 4 hours (4h), and 6 hours (6h) post-exercise in heparin vacutainer tubes. Peripheral blood mononuclear cells (PBMC) were isolated using Ficoll-Paque PLUS density gradient centrifugation. Total T cells were purified from washed PBMC by E-rosetting. T cell proliferation was analyzed in response to co-stimulation through CD3+CD28 using plate-bound antibodies, or phytohaemagglutinin (PHA) treatment, or no simulation. Cells were incubated for 6 days at 37˚C in a humidified incubator with 5% CO2 and then analyzed by flow cytometry. Cells were analyzed by flow cytometry using anti-CD3-APC, and anti-CD152-PE antibodies immediately after CD3+ T cell isolation (0 h) and following 6 d in culture using an Accuri C6 flow cytometer.

SECONDARY OUTCOMES:
Catecholamines (hormones) | 6.5 hours
  Blood will be collected in a vial containing EDTA (6 ml) for analysis of catecholamines. Plasma for catecholamine (epinephrine and norepinephrine) analyses was obtained by centrifugation at 2000 g for 10 min at 4˚C. The supernatant was removed and stored at -80˚C until analysis. Catecholamine concentrations will be determined using BI-CAT ELISA kits and performed per the manufacturer's instructions. The samples were measured at 450 nm using a Synergy HT microplate reader. The blood samples will be obtained at the same time as for the primary outcomes (prior to and following exercise as well as one, four and six hours post-exercise.
Complete Blood Count | 6.5 hours
  Peripheral blood will be collected in a vial containing EDTA (6 ml) for analysis of complete blood counts (CBC). These vials will be sent to a commercial clinical laboratory (Quest Diagnostics) for the CBC measures. The blood samples will be obtained at the same time as for the primary outcomes (prior to and following exercise as well as one, four and six hours post-exercise).
Cortisol | 6.5 hours
  Blood will be collected in a vial containing EDTA (6 ml) for analysis of cortisol. These vials will be sent to a commercial clinical laboratory (Quest Diagnostics) for the cortisol measures. The blood samples will be obtained at the same time as for the primary outcomes (prior to and following exercise as well as one, four and six hours post-exercise).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas, Lawrence, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF
Time Frame: Until December 29, 2025

REFERENCES:
- [Derived] Siedlik J, Deckert J, Dunbar A, Bhatta A, Gigliotti N, Chan M, Benedict S, Bubak M, Vardiman J, Gallagher P. Acute high-intensity exercise enhances T cell proliferation compared to moderate-intensity exercise. Appl Physiol Nutr Metab. 2025 Jan 1;50:1-12. doi: 10.1139/apnm-2024-0420. PMID 39947139